CLINICAL TRIAL: NCT02887326
Title: Keratoconus - Biomarkers and Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: AUH-3828
Record Dates: First submitted 2016-08-29; First posted 2016-09-02 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2017-10

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tear fluid, saliva and blood.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- age 15-25 years: Ophthalmic examination, VA measure, contrast vision, pentacam measurement, Tear fluid, saliva and blood samples
- age 25-35 years: Ophthalmic examination, VA measure, contrast vision, pentacam measurement, Tear fluid, saliva and blood samples
- age 35-45 year: Ophthalmic examination, VA measure, contrast vision, pentacam measurement, Tear fluid, saliva and blood samples
- > age 45 year: Ophthalmic examination, VA measure, contrast vision, pentacam measurement, Tear fluid, saliva and blood samples

SUMMARY:
The biomarker study adds to our previous study on biomarkers in tear fluid. In this study the investigators examine wether the biomarker levels are in correlation with the disease level and duration of disease.

The questionnaire study focuses on the patients perspective. With a validated questionnaire fore keratoconus patient it examine the patients self.-evaluated visual challenges and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Keratoconus residint in the Central Denmark Region

Exclusion Criteria:

* Other eye diseases
* Ocular traumas.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with keratoconus residing in the Central Denmark Region
Sampling Method: Non-Probability Sample
Enrollment: 287 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Protein levels in tear fluid, saliva and blood(plasma) | fall 2018
Ranch analysis of questionnaire | fall 2018

IPD SHARING:
Plan to Share IPD: No